CLINICAL TRIAL: NCT05152134
Title: Mobile & Online-Based Interventions to Lessen Pain (MOBILE Relief) in People With Prescription Opioid Misuse
Brief Title: Mobile & Online-Based Interventions to Lessen Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Beth Darnall, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61643; K24DA053564 (NIH)
Record Dates: First submitted 2021-10-07; First posted 2021-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain; Opioid Misuse; Opioid Use Disorder
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowered Relief On Demand (Experimental): Empowered Relief On-Demand will include roughly 80 minutes of interactive and multimedia pain educational content that targets pain and stress self-regulation, pain medication misuse, a personalized plan for relief and an audio App for daily use.
  Interventions: Behavioral: Empowered Relief On-Demand
- Health Education (HE; "Living Better") (Placebo Comparator): The HE arm is an interactive digital general health education intervention called "Living Better" that is devoid of specific content on pain, psychological skills, and has no active strategies or worksheets.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Empowered Relief On-Demand — Tailored interactive digital health treatment for chronic pain
  Arms: Empowered Relief On Demand
Behavioral: Health Education — The HE digital intervention is roughly 65 minutes with content discussing pain and health topics generally; it is devoid of pain education, psychological skills, and has no active strategies, worksheets, or supportive tools.
  Arms: Health Education (HE; "Living Better")

SUMMARY:
The investigators will implement an international 2-arm online pragmatic feasibility randomized controlled trial (RCT) of a digital pain relief skills intervention "Empowered Relief: On-Demand" to reduce pain metrics, opioid craving, and opioid misuse. They will compare Empowered Relief to a no-skills digital health education ("Living Better") intervention in community-based individuals with comorbid chronic pain and prescription opioid misuse (N=220). Completion of the brief post-treatment survey is a binary measure of treatment engagement; treatment feasibility and appraisal are assessed with three items (satisfaction, perceived utility, and likelihood to use skills learned). Electronic surveys will measure opioid misuse behaviors, craving, and use; and pain intensity and psychological status at: baseline, immediately post-treatment; at post-treatment weeks 1 and 2; and months 1, 2, and 3.

DETAILED DESCRIPTION:
Most people who misuse prescription opioids report doing so for pain relief. This study will investigate a digital intervention for people with comorbid chronic pain and opioid misuse.

The intervention, Empowered Relief On-Demand, will include roughly 80 minutes of interactive digital pain education and pain management skills content with multimedia features and an App. The investigators will conduct a fully online 2-arm RCT of digital Empowered Relief in a national sample of people with comorbid chronic pain and opioid misuse compared to a digital health education control (HE).

The investigators will implement The MOBILE Relief Study, an international (United States, Canada, United Kingdom, and Australia) 2-arm online feasibility RCT of Empowered Relief to reduce pain intensity, pain interference, pain-related distress (pain outcomes) and opioid outcomes (opioid craving and misuse) in people with prescription opioid misuse and chronic pain. They will compare Empowered Relief On Demand to an interactive digital health education (HE) intervention that is devoid of pain management skills ("Living Better") in community-based individuals with comorbid chronic pain and prescription opioid misuse (N=220). Completion of the brief post-treatment survey (received immediately following treatment completion) is a binary measure of treatment engagement; treatment feasibility and appraisal are assessed with five items (overall satisfaction with treatment, ease of understanding, relevance, perceived utility, and likelihood to use skills learned). Electronic surveys will measure opioid misuse behaviors, craving, and use; and pain intensity and psychological status at: baseline, and months 1, 2, and 3. At post-treatment weeks 1 and 2, electronic surveys will measure opioid craving, pain intensity, pain catastrophizing (distress), and pain interference.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 years of age or older
* Chronic non-cancer pain (at least 6 months in duration)
* Average pain intensity of at least 3 on the PROMIS SFV1.0 Pain Intensity 1a
* Daily prescription opioid use (at least 10 morphine milliequivalent daily dose; MEDD) for at least 3 months
* Opioid misuse (at least 6 on the Current Opioid Misuse Measure; COMM)
* English fluency
* Internet access

Exclusion Criteria:

* Gross cognitive impairment
* Inability to complete study electronic surveys
* Cannot currently be enrolled in a study or trial with Empowered Relief as a treatment/intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | baseline
  One validated item assessing average pain intensity for the past 7 days (0= "no pain" to 10= "worst pain imaginable").
Pain intensity | post-treatment week 1
  One validated item assessing average pain intensity for the past 7 days (0= "no pain" to 10= "worst pain imaginable").
Pain intensity | post-treatment week 2
  One validated item assessing average pain intensity for the past 7 days (0= "no pain" to 10= "worst pain imaginable").
Pain intensity | post-treatment month 1 (Multi-Primary Endpoint)
  One validated item assessing average pain intensity for the past 7 days (0= "no pain" to 10= "worst pain imaginable").
Pain intensity | post-treatment month 2
  One validated item assessing average pain intensity for the past 7 days (0= "no pain" to 10= "worst pain imaginable").
Pain intensity | post-treatment month 3
  One validated item assessing average pain intensity for the past 7 days (0= "no pain" to 10= "worst pain imaginable").
Pain catastrophizing | baseline
  A 13-item scale used to quantify an individual's pain experience (5 point scale where 0 = "Not at all" and 4 = "All the time"). Scores range from 0-52 with higher scores indicating higher levels of pain catastrophizing.
Pain catastrophizing | post-treatment week 1
  A brief 4-item scale used to quantify an individual's pain experience (5 point scale where 0 = "Not at all" and 4 = "All the time"). Scores range from 0-16 with higher scores indicating higher levels of pain catastrophizing.
Pain catastrophizing | post-treatment week 2
  A brief 4-item scale used to quantify an individual's pain experience (5 point scale where 0 = "Not at all" and 4 = "All the time"). Scores range from 0-16 with higher scores indicating higher levels of pain catastrophizing.
Pain catastrophizing | post-treatment month 1 (Multi-Primary Endpoint)
  A 13-item scale used to quantify an individual's pain experience (5 point scale where 0 = "Not at all" and 4 = "All the time"). Scores range from 0-52 with higher scores indicating higher levels of pain catastrophizing.
Pain catastrophizing | post-treatment month 2
  A 13-item scale used to quantify an individual's pain experience (5 point scale where 0 = "Not at all" and 4 = "All the time"). Scores range from 0-52 with higher scores indicating higher levels of pain catastrophizing.
Pain catastrophizing | post-treatment months 3
  A 13-item scale used to quantify an individual's pain experience (5 point scale where 0 = "Not at all" and 4 = "All the time"). Scores range from 0-52 with higher scores indicating higher levels of pain catastrophizing.
Pain interference | baseline
  6 items assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" with higher scores representing a greater degree of pain interference.
Pain interference | post-treatment week 1
  6 items assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" with higher scores representing a greater degree of pain interference.
Pain interference | post-treatment week 2
  6 items assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" with higher scores representing a greater degree of pain interference.
Pain interference | post-treatment month 1 (Multi-Primary Endpoint)
  6 items assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" with higher scores representing a greater degree of pain interference.
Pain interference | post-treatment month 2
  6 items assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" with higher scores representing a greater degree of pain interference.
Pain interference | post-treatment month 3
  6 items assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" with higher scores representing a greater degree of pain interference.
Current prescription opioid misuse | baseline
  17 items assessing opioid misuse thoughts and behaviors over the past 30 days. Four point response scale (0 = "never" to 4 = "very often") with higher scores representing more opioid misuse.
Current prescription opioid misuse | post-treatment month 1 (Primary Endpoint)
  17 items assessing opioid misuse thoughts and behaviors over the past 30 days. Four point response scale (0 = "never" to 4 = "very often") with higher scores representing more opioid misuse.
Current prescription opioid misuse | post-treatment month 2
  17 items assessing opioid misuse thoughts and behaviors over the past 30 days. Four point response scale (0 = "never" to 4 = "very often") with higher scores representing more opioid misuse.
Current prescription opioid misuse | post-treatment month 3 (Secondary Endpoint)
  17 items assessing opioid misuse thoughts and behaviors over the past 30 days. Four point response scale (0 = "never" to 4 = "very often") with higher scores representing more opioid misuse.
Opioid craving | baseline
  1 item asking participants to indicate how much opioid craving they have experienced over the past week (0 = "no craving" to 10 = "strongest craving ever").
Opioid craving | post-treatment week 1
  1 item asking participants to indicate how much opioid craving they have experienced over the past week (0 = "no craving" to 10 = "strongest craving ever").
Opioid craving | post-treatment week 2
  1 item asking participants to indicate how much opioid craving they have experienced over the past week (0 = "no craving" to 10 = "strongest craving ever").
Opioid craving | post-treatment month 1 (Primary Endpoint)
  1 item asking participants to indicate how much opioid craving they have experienced over the past week (0 = "no craving" to 10 = "strongest craving ever").
Opioid craving | post-treatment month 2
  1 item asking participants to indicate how much opioid craving they have experienced over the past week (0 = "no craving" to 10 = "strongest craving ever").
Opioid craving | post-treatment months 3 (Secondary Endpoint)
  1 item asking participants to indicate how much opioid craving they have experienced over the past week (0 = "no craving" to 10 = "strongest craving ever").
Opioid use | Baseline to post-treatment month 3
  Percent reduction (0-100%) of self-reported prescribed Morphine Equivalent Daily Dose (MEDD).
Treatment engagement | Immediately post-treatment (Primary Outcome)
  Proportion of participants in both study arms that complete the brief treatment appraisal survey administered immediately after treatment
Treatment appraisal | Immediately post-treatment (Primary Outcome)
  5 items assess satisfaction and perceived utility of assigned treatment (7-point scale where 0 = "not at all satisfied" to 6 = "extremely satisfied"). Higher scores indicate higher satisfaction with the assigned treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edwards KA, Palenski P, Perez L, You DS, Ziadni MS, Jung C, Adair E, Tian L, Mackey SC, Darnall BD. Protocol for a randomised trial of a self-directed digital pain management intervention (Empowered Relief) tailored to adults with chronic pain and prescription opioid misuse/disorder: the MOBILE Relief study. BMJ Open. 2024 Aug 9;14(8):e086889. doi: 10.1136/bmjopen-2024-086889. PMID 39122392